CLINICAL TRIAL: NCT01035515
Title: A Single-Center, Randomized, Placebo-Controlled, Double-Blind, Crossover Study to Evaluate the Cardiovascular Effects of Single Doses of Oral BIIB014 in Healthy Volunteers
Brief Title: BIIB014 Cardiovascular Monitoring Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Biogen Idec Study MD, Biogen Idec
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 204HV102
Record Dates: First submitted 2009-12-17; First posted 2009-12-18 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2010-06

CONDITIONS: Healthy
Keywords: Healthy subjects
MeSH Terms: interventions — 3-(4-amino-3-methylbenzyl)-7-(2-furyl)-3H-(1,2,3)triazolo(4,5-d)pyrimidine-5-amine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Arm One (Experimental): Arm 1 of 6 cross-over arms
  Interventions: Drug: Placebo; Drug: BIIB014 50mg; Drug: BIIB014 100mg
- Arm Two (Experimental): Arm 2 of 6 cross-over arms
  Interventions: Drug: Placebo; Drug: BIIB014 50mg; Drug: BIIB014 100mg
- Arm Three (Experimental): Arm 3 of 6 cross-over arms
  Interventions: Drug: Placebo; Drug: BIIB014 50mg; Drug: BIIB014 100mg
- Arm Four (Experimental): Arm 4 of 6 cross-over arms
  Interventions: Drug: Placebo; Drug: BIIB014 50mg; Drug: BIIB014 100mg
- Arm Five (Experimental): Arm 5 of 6 cross-over arms
  Interventions: Drug: Placebo; Drug: BIIB014 50mg; Drug: BIIB014 100mg
- Arm Six (Experimental): Arm 1 of 6 cross-over arms
  Interventions: Drug: Placebo; Drug: BIIB014 50mg; Drug: BIIB014 100mg

INTERVENTIONS:
Drug: Placebo — Single dose oral capsule placebo comparator
Drug: BIIB014 50mg — Single dose oral capsule 50mg BIIB014
Drug: BIIB014 100mg — Single dose oral capsule 100mg BIIB014

SUMMARY:
The study will examine the effects of a single dose of BIIB014 on blood pressure and haemodynamic variables in healthy volunteers over 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects
* Between the ages of 18 and 50, inclusive.
* Must have a body mass index (BMI) between 19 kg/m2 and 30 kg/m2, inclusive

Exclusion Criteria:

* Clinically significant abnormalities (as determined by the Investigator)
* Other unspecified reason that would make the subject unsuitable for enrollment (as determined by the Investigator)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-12; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Supine Blood pressure | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Quintiles Inc, Overland Park, Kansas, United States